CLINICAL TRIAL: NCT00100347
Title: A Phase 1 Dose Escalation Safety/Tolerance Study of PPI-2458 in Subjects With Non-Hodgkin's Lymphoma and Solid Tumors
Brief Title: Safety/Tolerance Study of PPI-2458 in Subjects With Non-Hodgkin's Lymphoma and Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: terminated due to corporate transaction.
Sponsor: PRAECIS Pharmaceuticals Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2458-04-01
Record Dates: First submitted 2004-12-29; First posted 2004-12-30 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Non-Hodgkin's Lymphoma,; Solid Tumors
Keywords: non-Hodgkin lymphoma; non-Hodgkin's lymphoma; NHL; MetAP2; Solid Tumors
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — PPI 2458

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PPI-2458

SUMMARY:
The purpose of this multi-center, open-label, escalating dose study is to assess the safety and tolerability of PPI-2458 in subjects with Non-Hodgkin's Lymphoma (NHL)and solid tumors. Subjects will be treated every other day (QOD) with PPI-2458 while being monitored closely for adverse events.

DETAILED DESCRIPTION:
The study will first determine the dose level that maximally inhibits MetAP2 in white blood cells (WBC). Once this dose level is reached, the study will proceed into the next cohort (dose level) to investigate the dose level that maximally inhibits MetAP2 in tumor tissue biopsies. Free MetAP2 levels (WBC and/or tumor tissue) will be analyzed during the first cycle (28 days) of treatment. Cohorts are expected to enroll every two cycles until the maximum tolerated dose (MTD)is determined.

After the Initial Treatment Phase of two treatment cycles of PPI-2458, subjects may continue into a Continuous Treatment Phase at the discretion of the Investigator. In order to be eligible for the Continuous Treatment Phase of the protocol, subjects must have received some benefit (e.g., stable disease) as assessed by the Investigator within the Initial Treatment Phase and must continue to meet inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the ability to understand the requirements of the study, provide written informed consent, and abide by the requirements of the study
* Male or female ≥ 18 years of age
* NHL subjects must have histologically confirmed (by the investigator) diffuse large B cell lymphoma (DLBCL) or follicular lymphoma (FL)- Grade I-III non-Hodgkin's lymphoma (including transformed subjects) with confirmed failure of prior treatment, defined as: a) Progression following other chemotherapy regimens, radiation therapy, monoclonal antibody therapy, or high dose therapy and autologous stem cell transplantation OR b) Not a candidate for or unwilling to undergo high dose therapy with autologous cell transplantation for DLBCL subjects, OR c) Received at least two previous treatment regimens for FL or relapsed, or progressed, while on or following cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) or anthracycline-based regimen for DLBCL subjects Solid tumor subjects must have histologically or cytologically confirmed solid tumor that is either measurable or evaluable and refractory to standard treatment or fow which no curative treatment exists.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 or Karnofsky performance status of 60 - 100%
* Life expectancy ≥ 2 months
* Laboratory values: *Absolute neutrophil count (ANC) ≥ 1,500/mm3; *Platelets ≥ 90,000/mm3; *Aspartate aminotransferase (AST) ≤ 2x upper limit of normal (ULN); *Alanine aminotransferase (ALT) ≤ 2x ULN; *Total bilirubin ≤ 1.5x ULN; *Serum creatinine < 1.5x ULN
* ≥ 3 weeks since chemotherapy, radiation therapy, monoclonal antibody therapy (e.g. rituximab, etc.) or major surgery, and ≥ 12 weeks since radioimmune therapy
* Results of the two baseline neurodiagnostic nerve conduction velocities (taken at least one week apart) may not vary more than 10%. Response must be well formed and clearl measurable, as judged by the electrophysiology core lab
* Women of childbearing potential must not be breastfeeding or lactating and must have a negative serum pregnancy test within 72 hours of starting the study
* Fertile males and females of child-bearing potential must practice medically acceptable contraception
* Confirmed HIV negative
* Tumor tissue cohorts only: Subjects must have accessible tumor tissue and be willing to undergo tumor tissue biopsies (2-4 core biopsies)
* For subjects entering Continuous Treatment Phase: Subjects must have received some benefit from the Initial Treatment Phase of PPI-2458 treatment (e.g., stable disease) as assessed by the Investigator.

Exclusion Criteria:

* Active central nervous system (CNS) lymphoma or brain metastases as evidenced by clinical symptoms or by computed tomography (CT) scan or magnetic resonance imaging (MRI), or progression from prior imaging
* A neuropathy ≥ Grade 2
* Baseline nerve conduction velocities, which vary by more than 10% and are inconsistent and/or poorly formed, as judged by the electrophysiology core lab
* Requirement for corticosteroids
* History of allogeneic stem cell transplantation
* History of seizures
* Active colitis, peptic ulcers, or Irritable Bowel Disease
* Any uncontrolled serious medical or psychiatric illness
* Electrocardiogram (ECG) showing clinically significant atrial or ventricular arrhythmias, 2nd degree or 3rd degree heart block or prolonged QTc interval > 480 msec
* Subjects taking any drug that is a known clinically relevant inhibitor or inducer of cytochrome P450 3A4.
* Has received an investigational drug within 21 days of study entry, is currently participating in another study, or is planning to participate in another study during this clinical trial
* Receiving ongoing pharmacological or radiological treatments for NHL
* History of mucositis, not related to prior NHL therapy, > Grade 1 within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-12; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety will be determined by clinical adverse events, laboratory abnormalities, withdrawals due to adverse events, and drug-related neurotoxicities.

SECONDARY OUTCOMES:
Pharmacokinetic assessment of PPI-2458
Pharmacodynamic assessment of PPI-2458

CONTACTS AND LOCATIONS:
Overall Officials: Paul Eder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - Universtiy of Maryland Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of New Mexico, Albuquerque, New Mexico
  - Columbia University Medical Center, New York, New York
  - University of Texas, M.D. Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia